CLINICAL TRIAL: NCT06356389
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase Ib/II Clinical Trial to Evaluate the Safety, Tolerance and Pharmacokinetic Characteristics of JX11502MA Capsules in Patients With Schizophrenia.
Brief Title: A Clinical Trial to Evaluate Safety, Tolerance and Pharmacokinetics of JX11502MA Capsule in Patients With Schizophrenia.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang Jingxin Pharmaceutical Co., Ltd. (Industry)
Collaborators: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JX11502MA-Ib-II
Record Dates: First submitted 2023-02-20; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JX11502MA (Experimental): JX11502MA 1.5 mg; JX11502MA 3 mg; JX11502MA 6 mg;
  Interventions: Drug: JX11502MA
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JX11502MA — Oral capsule
  Arms: JX11502MA
Drug: Placebo — Oral capsule
  Arms: Placebo

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled, dose-increasing phase Ib/II clinical trial to evaluate the safety, tolerance and pharmacokinetic characteristics of JX11502MA capsules administered multiple times in patients with schizophrenia

DETAILED DESCRIPTION:
This study adopts a multi-center, randomized, double-blind, dose-increasing, parallel-control titration drug delivery study design.

Preset three dose groups (S1, S2, S3), low, medium and high, with target doses of 1.5mg, 3mg and 6mg respectively. Each dose group included 20 subjects (16 patients received the test drug and 4 patients received placebo). During the test, observe the safety and tolerance of the subjects, and collect PK blood samples.

Schizophrenic patients who met the inclusion criteria after screening and evaluation were randomly enrolled on the baseline day. On the first administration day, all dose groups took 1.5mg as the starting dose. Each subject should closely observe the tolerance and safety within 24 hours after the first administration. Only when the investigator evaluated it as tolerable, can the subsequent multiple administration be continued.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of signing the informed consent form, 18 years old ≤ 55 years old, male and female are not limited;
2. 18.5kg/m2 ≤ body mass index (BMI) ≤ 30kg/m2, and male weight ≥ 50kg, female weight ≥ 45kg;
3. Subjects were diagnosed as schizophrenia according to DSM-5 diagnostic criteria;
4. Subjects are currently taking second-generation antipsychotics (≤ 2 kinds, except for clozapine and long-acting preparations), the dose does not exceed the maximum dose specified in the instructions, and the dose and frequency of administration are basically stable in the past 2 weeks; Or currently useless drugs but taking second-generation antipsychotic drugs in the past ≥ 2 weeks;
5. The total score of the PANSS scale in the screening period is less than 90 points, of which the following items are scored ≤ 4 points (such as P4, P6, P7, G2, G4, G8, G14);
6. Female and male subjects of childbearing age and their spouses need to be able to effectively contraception (medically approved contraceptives, such as intrauterine devices, contraceptives or condoms) during the study medication period and within 6 months after the end of medication;
7. The subjects and their guardians fully understand the purpose and requirements of the trial, voluntarily participate in the clinical trial and sign the written informed consent form, and are willing to complete the whole trial process according to the trial requirements.

Exclusion Criteria:

1. Patients who meet the DSM-5 diagnostic criteria for other mental diseases;
2. Use long-acting antipsychotic drugs within 6 months before the first administration;
3. He received electric shock treatment and transcranial magnetic stimulation (rTMS) within 3 months before screening;
4. The answer to question 4 or 5 of the Columbia Suicide Scale (C-SSRS) suicide ideation in the screening period is "yes", or the person who has obvious suicide tendency at present or in the past 12 months, or the researcher believes that there is a risk of suicide and violence based on the clinical evaluation of the researcher;
5. Those with abnormal physical examination or vital signs in screening period and significant clinical significance;
6. The laboratory examination during the screening period was abnormal, and the researcher determined that it was of obvious clinical significance, such as: liver: glutamate aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 1.5 times the upper limit of the normal value; Kidney: creatinine (Cr)>upper limit of normal value;
7. The increase of prolactin in the screening period is judged by the researcher to have obvious clinical significance (such as amenorrhea, breast development and other clinical symptoms);
8. During the screening period, the subjects' systolic blood pressure was<90mmHg or>140mmHg, and their diastolic blood pressure was<60mmHg or>90mmHg;
9. Diabetes patients with poor control (fasting blood glucose ≥ 10mmol/L), or are using insulin to treat diabetes, or initially diagnosed as type 2 diabetes at screening;
10. Those with QTc interval>450ms (male) or 470ms (female) in the screening period, or with family history of long QT interval syndrome, or with cardiac insufficiency, serious arrhythmia or ischemic heart disease and requiring drug treatment, have congenital heart disease, serious organic heart disease or a history of this disease;
11. Those with epilepsy and other convulsive diseases (except for febrile convulsion);
12. Those with serious or unstable cardiovascular, respiratory, liver, kidney, blood, endocrine, nervous system or other system diseases;
13. Smokers who smoke more than 10 cigarettes or the same amount of cigarettes per day within 3 months before screening;
14. Those who drink alcohol within 6 months before screening and have an average weekly alcohol intake of more than 14 units (1 unit=285 mL of beer or 25 mL of spirits or 150 mL of wine) or who have positive alcohol breath test;
15. Those who have a history of drug and drug abuse within one year before screening, or who are positive for urine drug screening (excluding benzodiazepine);
16. Subjects who may be allergic to any component of this drug or its analogues;
17. HIV antibody, HBsAg, HCV antibody or syphilis serological test result is positive;
18. There is obvious history of blood loss, blood donation or blood loss ≥ 200mL within 3 months before screening;
19. Those who have been enrolled in other clinical trials or are participating in clinical trials within 3 months before screening;
20. Pregnant or lactating women;
21. The researcher thinks it is not suitable to participate in this test.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Day1 to Day 28
  The number and percentage of participants with TEAEs will be determined

SECONDARY OUTCOMES:
Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Day 28 | Day1 to Day 28
  The PANSS rating form contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. For negative symptoms in schizophrenia, participants are rated from 1 to 7 on each symptom scale, with a minimum score of 7 and a maximum score of 49. A decrease in PANSS total score correlates with an improvement in schizophrenia symptoms.
Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Positive Score at Day 28 | Day1 to Day 28
  The PANSS rating form contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. For positive symptoms in schizophrenia, participants are rated from 1 to 7 on each symptom scale, with a minimum score of 7 and a maximum score of 49. A decrease in PANSS total score correlates with an improvement in schizophrenia symptoms.
Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Negative Score at Day 28 | Day1 to Day 28
  The PANSS rating form contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. For negative symptoms in schizophrenia, participants are rated from 1 to 7 on each symptom scale, with a minimum score of 7 and a maximum score of 49. A decrease in PANSS total score correlates with an improvement in schizophrenia symptoms.
Change From Baseline in Clinical Global Impression - Severity (CGI-S) Score at Day 28 | Day1 to Day 28
  The CGI-S modified asked the clinician 1 question: "Considering your total clinical experience, how mentally ill is the participant at this time?" The clinician's answer rated on the following 7-point scale: 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill participants.
Tmax | Day1 to Day 28
  Peak time
Css_min | Day1 to Day 28
  Steady-state trough concentration
Css_max | Day1 to Day 28
  Steady-state peak concentration
Css_av | Day1 to Day 28
  Mean steady-state blood drug concentration
AUC0-t,ss | Day1 to Day 28
  Area under the plasma concentration-time curve from the last dose to the last measurable concentration time point
AUC0-∞,ss | Day1 to Day 28
  Extrapolated area under the plasma concentration-time curve from the last dose to infinity
AUCtau,ss | Day1 to Day 28
  Area under the plasma concentration-time curve within one dosing interval at steady state
t1/2 | Day1 to Day 28
  Elimination half-life

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No